CLINICAL TRIAL: NCT02728843
Title: A Dose-Ranging Study of the Efficacy, Safety, and Pharmacokinetics of Deferiprone Delayed Release Tablets in Patients With Parkinson's Disease
Brief Title: Study of Parkinson's Early Stage With Deferiprone
Acronym: SKY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Organization: Chiesi Canada Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LA48-0215
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deferiprone
MeSH Terms: conditions — Parkinson Disease | interventions — Deferiprone; Isoflurophate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo tablets had the same appearance as the deferiprone tablets, and within each dosing cohort, all participants took the same number of tablets at each dose.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Deferiprone 300 mg (Experimental): One-half of a 600 mg tablet of deferiprone twice a day, for a total daily dosage of 600 mg
  Interventions: Drug: Deferiprone
- Deferiprone 600 mg (Experimental): One 600 mg tablet of deferiprone twice a day, for a total daily dosage of 1200 mg
  Interventions: Drug: Deferiprone
- Deferiprone 900 mg (Experimental): One and a half 600 mg tablets of deferiprone twice a day, for a total daily dosage of 1800 mg
  Interventions: Drug: Deferiprone
- Deferiprone 1200 mg (Experimental): Two 600 mg tablets of deferiprone twice a day, for a total daily dosage of 2400 mg
  Interventions: Drug: Deferiprone
- Placebo (Placebo Comparator): Depending on dosage cohort, either one half-tablet, one tablet, one and a half tablets, or two tablets of placebo, twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferiprone — 600 mg tablets
  Other Names: DFP
  Arms: Deferiprone 1200 mg; Deferiprone 300 mg; Deferiprone 600 mg; Deferiprone 900 mg
Drug: Placebo — Tablets that match the deferiprone tablets in appearance
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the effects of deferiprone, an iron-chelating drug, in patients with Parkinson's disease. Participants will be randomized to receive one of four different dosages of deferiprone or placebo, and will take the assigned study product twice a day for nine months.

DETAILED DESCRIPTION:
This study will enroll 140 patients who have been diagnosed with Parkinson's disease within the last 3 years and are currently taking antiparkinsonian medication. There are four dosage cohorts, with patients in each cohort receiving either deferiprone tablets or placebo. At the baseline visit, participants will be randomized to a dosage cohort and to either active product or placebo within that cohort, and will take the assigned study product twice-daily for 9 months. They will come back to the study site for assessments at Months 1, 2, 3, 4, 5, 6, and 9, and will need to have their blood count checked weekly, at either the study site or a local laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 to < 80 years
* Body weight ≥60 kg but ≤100 kg
* Parkinson's disease diagnosed
* Absolute neutrophil count (ANC) ≥1.5 x 10^9/L (≥1.0 x 10^9/L for Black population) at screening
* On a stable dose for at least 3 months prior to the screening visit of any of the following treatments at an L-dopa equivalent daily dose of up to 600 mg:
* Dopaminergic agonist alone
* L-dopa alone
* Combination therapy with dopaminergic agonist and L-dopa
* Rasagiline
* At an early stage of the disease, without motor fluctuations and/or L-dopa-induced dyskinesia

Exclusion Criteria:

* Diagnosis of Parkinson's disease more than 3 years prior to screening visit
* Hoehn and Yahr stage ≥ 3
* Atypical or secondary Parkinsonism without dopa-sensitivity (e.g., vascular parkinsonism, supranuclear palsy, multisystem atrophy)
* Progressing Axis I psychiatric disorders (psychosis, hallucinations, compulsive disorders, substance addiction, bipolar disorder, severe depression, anxiety) as assessed in a semi-structured interview in accordance with the Diagnostic and Statistical Manual of Mental Disorders
* Not stabilized in terms of the current antiparkinsonian therapeutic regimen: already requires dose adaptation and/or is likely to require any change in dopamine therapy over the duration of the trial
* Current treatment with bromocriptine
* Current treatment with any antiparkinsonian drug other than those listed in the inclusion criteria
* Current treatment with coenzyme Q10 or idebenone. (Patients who are on these medications but stop taking them at least 2 weeks prior to baseline may be enrolled.)
* Current use of a Deep Brain Stimulation (DBS) system. (Patients who previously had a DBS system but have had it removed may be enrolled.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, Principal Investigator — Hospitalier Régional Universitaire de Lille
Locations (20):
- Toronto Western Hospital, Toronto, Ontario, Canada
- France (10):
  - CHU de Bordeaux, Centre Expert Parkinson, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Régional Universitaire de Lille, Hôpital Roger Salengro, Lille
  - CHU Dupuytren, Limoges
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU Pontchaillou, Rennes
  - CHU Charles Nicoll - Rouen, Rouen
  - Hôpitaux Universitaires de Strasbourg, Hôpital de Hautepierre, Strasbourg
  - CHU Purpan, Hôpital Pierre Paul Riquet, Toulouse
- Germany (4):
  - Heinriche-Heine Universität Düsseldorf, Düsseldorf
  - UKSH Campus Kiel, Neurologie, Kiel
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Klinikum rechts der Isar, Munich
- United Kingdom (5):
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - Fairfield General Hospital, Bury
  - Charing Cross Hospital, London
  - Newcastle Clinical Ageing Research Unit, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devos D, Rascol O, Meissner WG, Foubert-Samier A, Lewis S, Tranchant C, Anheim M, Maltete D, Remy P, Eggert K, Pape H, Geny C, Couratier P, Carroll C, Sheridan R, Burn D, Pavese N, Raw J, Berg D, Suchowersky O, Kalia LV, Evans A, Drapier S, Danaila T, Schnitzler A, Corvol JC, Defer G, Temin NT, Fradette C, Tricta F, Moreau C; a Parkinson's disease study group. Therapeutic modalities of deferiprone in Parkinson's disease: SKY and EMBARK studies. J Parkinsons Dis. 2025 Feb;15(1):72-86. doi: 10.1177/1877718X241300295. Epub 2024 Dec 27. PMID 39973479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Started | 28 | 28 | 28 | 28 | 28
Completed | 25 | 23 | 20 | 22 | 23
Not Completed | 3 | 5 | 8 | 6 | 5
Not completed — Adverse Event | 0 | 2 | 3 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 4 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Use of rescue medication | 0 | 2 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Only patients in the Intent to Treat (ITT) population are presented. The ITT population was defined as all randomized patients who received at least one dose of study drug and had a baseline and at least one post-baseline efficacy assessment for the primary endpoint.
Groups:
- 300 mg: Patients took 300 mg deferiprone twice daily, for a total daily dosage of 600 mg
- 600 mg: Patients took 600 mg deferiprone twice daily, for a total daily dosage of 1200 mg
- 900 mg: Patients took 900 mg deferiprone twice daily, for a total daily dosage of 1800 mg
- 1200 mg: Patients took 1200 mg deferiprone twice daily, for a total daily dosage of 2400 mg
- Placebo: Depending on which dosage cohort they were in, patients took a number of placebo tablets that matched the number of tablets taken by patients receiving active product
- Total: Total of all reporting groups
Arm/Group | 300 mg | 600 mg | 900 mg | 1200 mg | Placebo | Total
Number analyzed (Participants) | 27 | 26 | 25 | 28 | 27 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.7) | 63.2 (8.5) | 59.8 (10.2) | 60.3 (8.7) | 61.9 (9.2) | 61.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 6 | 15 | 6 | 43
  Male | 17 | 20 | 19 | 13 | 21 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 26 | 26 | 25 | 26 | 26 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 27 | 25 | 25 | 26 | 27 | 130
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 1 | 1 | 1 | 3
  United Kingdom | 6 | 4 | 3 | 6 | 6 | 25
  France | 17 | 19 | 18 | 21 | 18 | 93
  Germany | 4 | 3 | 3 | 0 | 2 | 12
MDS-UPDRS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is used to follow the longitudinal course of Parkinson's disease. It contains 4 parts. Each item has a rating of 0-4: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). The total score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability.
  units on a scale | 29.7 (11.6) | 31.1 (13.3) | 29.8 (12.3) | 24.5 (10.7) | 27.4 (12.3) | 28.4 (12.1)
MDS-UPDRS Part I [Mean (Standard Deviation); unit: units on a scale] — Part I of the MDS-UPDRS is the subscale that evaluates mentation, behavior, and mood. Scores range from 0 (best) to 52 (worst).
  units on a scale | 6.2 (4.1) | 5.7 (3.0) | 5.9 (3.4) | 5.3 (2.4) | 5.0 (3.1) | 5.6 (3.2)
MDS-UPDRS Part II [Mean (Standard Deviation); unit: units on a scale] — Part II of the MDS-UPDRS is the subscale for motor experiences of daily living. Scores range from 0 (best) to 52 (worst).
  units on a scale | 4.1 (3.5) | 5.8 (3.9) | 5.7 (5.0) | 3.9 (3.1) | 6.1 (4.0) | 5.1 (4.0)
MDS-UPDRS Part III [Mean (Standard Deviation); unit: units on a scale] — Part III of the MDS-UPDRS is the subscale for motor examination. Scores range from 0 (best) to 132 (worst).
  units on a scale | 19.1 (7.8) | 19.4 (10.4) | 18.1 (7.8) | 15.1 (8.5) | 16.3 (9.1) | 17.6 (8.8)
MDS-UPDRS Part II/Part III [Mean (Standard Deviation); unit: units on a scale] — The combined score from the Part II subscale (motor experiences of daily living) and the Part III subscale (motor examination) of the MDS-UPDRS. For Part II, scores can range from 0 (best) to 52 (worst), and for Part III, they can range from 0 (best) to 132 (worst). Hence, the combined score can range from 0 (best) to 184 (worst).
  units on a scale | 23.2 (10.1) | 25.2 (12.4) | 23.8 (10.8) | 19.1 (9.9) | 22.4 (10.6) | 22.7 (10.8)
MDS-UPDRS Part IV [Mean (Standard Deviation); unit: units on a scale] — Part IV of the MDS-UPDRS is the subscale for motor complications. Scores range from 0 (best) to 24 (worst).
  units on a scale | 0.2 (0.8) | 0.2 (0.8) | 0.1 (0.6) | 0.2 (0.8) | 0.0 (0.2) | 0.2 (0.7)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) test is a rapid screening instrument for the detection of mild cognitive dysfunction. It is used to assess the following cognitive domains: short-term memory recall, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place. The total score on the MoCA can range from 0 (worst) to 30 (best).
  units on a scale | 27.7 (1.3) | 28.1 (1.7) | 27.3 (1.9) | 27.5 (2.0) | 27.1 (1.9) | 27.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on the Part III Subscale of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: Change from baseline to Month 9 in the score for the Part III subscale (motor examination) of the MDS-UPDRS. Scores on this subscale can range from 0 (best) to 132 (worst); hence, an increase would indicate progression of the disease and a decrease would indicate improvement. The change in score was calculated as least square means.
Time Frame: Nine months
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | 2.1 (1.4) | 4.2 (1.4) | -0.8 (1.5) | 3.9 (1.5) | 2.2 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 900 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

2. Secondary Outcome: Change in Total Score on the MDS-UPDRS
Description: Change from baseline to Month 9 in total score on the MDS-UPDRS. The total score can range from 0 (best) to 260 (worst); hence, an increase would indicate progression of the disease and a decrease would indicate improvement. The change in score was calculated as least square means.
Time Frame: Nine months
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | 4.1 (1.9) | 7.8 (1.9) | 0.5 (2.1) | 6.6 (2.1) | 5.9 (2.0)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 900 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

3. Secondary Outcome: Change in Score on the Part I Subscale of the MDS-UPDRS
Description: Change from baseline to Month 9 in the score for the Part I subscale (mentation, behavior, and mood) of the MDS-UPDRS. Scores on this subscale can range from 0 (best) to 52 (worst); hence, an increase would indicate progression of the disease and a decrease would indicate improvement. The change in score was calculated as least square means.
Time Frame: Nine months
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | 0.8 (0.7) | 1.0 (0.7) | 0.3 (0.7) | 0.3 (0.7) | 1.1 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 900 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

4. Secondary Outcome: Change in Score on the Part II Subscale of the MDS-UPDRS
Description: Change from baseline to Month 9 in the score for the Part II subscale (activities of daily living) of the MDS-UPDRS. Scores on this subscale can range from 0 (best) to 52 (worst); hence, an increase would indicate progression of the disease and a decrease would indicate improvement. The change in score was calculated as least square means.
Time Frame: Nine months
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | 1.1 (0.6) | 2.2 (0.6) | 0.6 (0.6) | 2.1 (0.6) | 1.8 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

5. Secondary Outcome: Change in Score in the Part IV Subscale of the MDS-UPDRS
Description: Change from baseline to Month 9 in the score for the Part IV subscale (motor complications) of the MDS-UPDRS. Scores on this subscale can range from 0 (best) to 24 (worst); hence, an increase would indicate progression of the disease and a decrease would indicate improvement. The change in score was calculated as least square means.
Time Frame: Nine months
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | -0.1 (0.2) | 0.2 (0.2) | 0.3 (0.2) | 0.2 (0.2) | 0.4 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 900 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

6. Secondary Outcome: Change in the Combined Scores From Parts II and III of the MDS-UPDRS
Description: Change from baseline to Month 9 in the combined score for the Part II subscale (motor experiences of daily living) and the Part III subscale (motor examination) of the MDS-UPDRS. The scales for these two parts range from 0 (best) to 52 (worst) and from 0 (best) to 132 (worst), respectively. Hence, the combined score can range from 0 (best) to 184 (worst), and an increase would indicate progression of the disease and a decrease would indicate improvement. The change in score is presented as least square means.
Time Frame: Nine months
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | 3.3 (1.6) | 6.5 (1.6) | -0.3 (1.7) | 6.0 (1.7) | 4.3 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 900 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

7. Secondary Outcome: Change in Score on the Montreal Cognitive Assessment (MoCA) Test
Description: Change from baseline to Month 9 in the score for overall cognitive function as assessed by the MoCA. The total score on the MoCA can range from 0 (worst) to 30 (best). Hence, a decrease in score would indicate progression of the disease and an increase would indicate improvement. The change in score is presented as least square means.
Time Frame: Nine months
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 25 | 28
Score on a scale | 1.1 (0.3) | 1.0 (0.3) | 0.9 (0.3) | 1.1 (0.3) | 1.4 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 300 mg vs Deferiprone 600 mg vs Deferiprone 900 mg vs Deferiprone 1200 mg; Test type: Superiority; p > 0.05, ANCOVA

8. Secondary Outcome: Safety of Deferiprone
Description: Number of subjects with adverse events
Time Frame: Nine months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
Participants | 26 | 25 | 23 | 25 | 25

9. Secondary Outcome: Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Blood samples for pharmacokinetics assessments were collected at baseline, and at pre-dose and specified time points up to 12 hours post-dose at the Month 3 visit. The maximum measured serum concentration (Cmax) at the Month 3 visit was determined for deferiprone and its main metabolite, deferiprone 3-O-glucuronide.
Time Frame: 4 hours
Population: Pharmacokinetics (PK) population: Included all patients who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 300 mg | 600 mg | 900 mg | 1200 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
μg/mL
  Serum deferiprone | 2.748 (0.781) | 3.459 (0.078) | 5.080 (2.614) | 7.942 (2.192)
  Serum deferiprone 3-O-glucuronide | 7.844 (0.936) | 12.419 (2.218) | 21.914 (8.309) | 32.632 (2.167)

10. Secondary Outcome: Tmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Blood samples for pharmacokinetics assessments were collected at baseline, and at pre-dose and specified time points up to 12 hours post-dose at the Month 3 visit. The time to maximum observed serum concentration (Tmax) at the Month 3 visit was determined for deferiprone and its main metabolite, deferiprone 3-O-glucuronide.
Time Frame: 4 hours
Population: Pharmacokinetics population: Included all patients who had sufficient PK data to derive at least one PK parameter.
Measure: Median (Full Range); unit: Hours
Arm/Group | 300 mg | 600 mg | 900 mg | 1200 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
Hours
  Serum deferiprone | 2.00 [1.67 to 2.33] | 2.17 [2.00 to 2.33] | 2.00 [0.58 to 2.67] | 1.67 [1.33 to 2.00]
  Serum deferiprone 3-O-glucuronide | 2.84 [2.33 to 3.00] | 3.25 [3.00 to 3.50] | 3.50 [2.67 to 3.58] | 2.50 [2.33 to 2.67]

11. Secondary Outcome: Area Under the Curve for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Blood samples for pharmacokinetics assessments were collected at baseline, and at pre-dose and specified time points up to 12 hours post-dose at the Month 3 visit. The total drug exposure, AUC0-∞ (area under the serum concentration time curve extrapolated to infinity) at the Month 3 visit was determined for deferiprone and its main metabolite, deferiprone 3-O-glucuronide.
Time Frame: 4 hours
Population: Pharmacokinetics population: Included all patients who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 300 mg | 600 mg | 900 mg | 1200 mg
Number analyzed (Participants) | 4 | 1 | 5 | 2
μg*h/mL
  Serum deferiprone | 8.358 (0.904) | 16.292 | 20.606 (8.742) | 26.328 (5.693)
  Serum deferiprone 3-O-glucuronide | 39.057 (7.820) | 62.679 | 121.128 (43.727) | 147.397 (6.502)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Placebo | Deferiprone 300 mg | Deferiprone 600 mg | Deferiprone 900 mg | Deferiprone 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/28 | 3/28 | 4/28 | 1/28
Other Adverse Events (participants affected / at risk) | 26/28 | 25/28 | 23/28 | 25/28 | 25/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Deferiprone 300 mg (N=28) | Deferiprone 600 mg (N=28) | Deferiprone 900 mg (N=28) | Deferiprone 1200 mg (N=28)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jealous delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Deferiprone 300 mg (N=28) | Deferiprone 600 mg (N=28) | Deferiprone 900 mg (N=28) | Deferiprone 1200 mg (N=28)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (4) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (2) | 2 (2) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5) | 2 (4) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 3 (4) | 2 (5) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 5 (8) | 2 (3) | 6 (8) | 4 (5)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (6)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (2) | 3 (3) | 2 (5) | 5 (6) | 4 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (4) | 2 (2) | 3 (4) | 2 (17) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood urine present (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 4 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 3 (4)
Akinesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 2 (3) | 2 (2) | 1 (2) | 3 (6)
Headache (Nervous system disorders) | 2 (6) | 6 (9) | 4 (4) | 5 (9) | 8 (29)
Parkinson's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 6 (8) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (2) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT02728843/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT02728843/SAP_001.pdf
  • Informed Consent Form (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT02728843/ICF_002.pdf